CLINICAL TRIAL: NCT00766987
Title: Ontario Provincial Registry Project for Cardiac Viability Assessment Using FDG PET
Brief Title: Cardiac FDG PET Viability Registry
Acronym: CADRE
Status: Completed | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Rob Beanlands, Robert S. Beanlands, MD, FRCPC, Chief of Cardiology, Ottawa Heart Institute Research Corporation
Other Study IDs: 2007437-01H; MOH-06374
Record Dates: First submitted 2008-10-02; First posted 2008-10-06 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure; Ischemic Heart Disease; Myocardial Dysfunction
Keywords: coronary artery disease; FDG PET viability imaging; morbidity and mortality; revascularization; resource utilization
MeSH Terms: conditions — Heart Failure; Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Positron Emission Tomography (PET) is a non-invasive, unique nuclear imaging technique that allows the evaluation of blood flow in the heart and provides information about the cell activity of specific organs such as the heart and brain. It also provides useful information for the management of patients with poor pumping function of the heart, heart failure, and coronary artery disease. A cardiac viability imaging looks at how the heart uses glucose (sugar) The imaging process determines areas of the heart that are alive (viable - using sugar) versus areas of the heart that are scar tissue (non-viable). F-18 fluorodeoxyglucose (FDG) is the radioactive substance used to determine myocardial viability. This nuclear imaging technique has been shown to be useful in directing management for patient care.

The Ministry of Health recognizes the clinical utility of FDG PET imaging for myocardial viability assessment and other cancer indications. Optimizing the potential advantages of FDG PET in Ontario, will require characterization of the patient population, referral patterns, upstream and downstream resource utilization and patient outcomes. Therefore, registry studies are being undertaken to provide specific information about the utility of PET in these clinical situations in Ontario. The proposed registry will facilitate monitoring of the implementation of this limited technology and allow continued evaluation of practice patterns and outcomes. The University of Ottawa Heart Institute is the coordinating centre for this project with PET centres in London, Hamilton and Toronto also participating.

The purpose of this study is to evaluate the utility of FDG PET viability imaging in the decision making process for patients with poor left ventricular function who may be candidates for revascularization and to study the downstream effect of the clinical management decisions. Patients meeting specific inclusion criteria will be eligible for this study.

DETAILED DESCRIPTION:
Heart failure from reduced left ventricular function is associated with significant morbidity and mortality and although there have been multiple trials involving medical and devices therapies that have shown improved survival, the overall mortality remains high. Therapeutic intervention studies involving transplantation and revascularization concluded that patients with viable myocardium can be revascularized but this approach is often not adopted because of high peri-operative morbidity and mortality.

Due to these factors there is a need for a better approach to define and select patients with severe ventricular dysfunction. FDG PET studies to date have consistently shown that patients with viable myocardium on FDG PET are at high risk for other cardiac events and death if they do not undergo timely revascularization. FDG PET viability data has had an impact on decision making in patients with severe left ventricular (LV) dysfunction and the benefits of early revascularization have been seen in patients with ischemic viable myocardium.

The accuracy of FDG PET to predict regional and global LV function recovery, its utility in decision making and ability to identify high risk patients have all been demonstrated. These findings all support a clinical role for FDG PET in assessing select patients with CAD and severe LV function. The Cardiac FDG PET Registry (CADRE) will provide specific information about the utility of PET in clinical situations. To our knowledge this is the largest multi-centre FDG PET myocardial viability registry. The registry will facilitate monitoring of and evaluation of practise patterns, upstream and downstream resource utilization (diagnostic imaging and revascularization) and outcomes as they relate to the severity of the abnormalities detected. The impact of FDG PET parameters on outcome measures will be compared to other clinical parameters. These findings will optimize the implementation of this technology in clinical practise in Ontario and further identify parameters that with FDG PET predict adverse outcomes for specific patient populations. The results of this registry will impact clinical practise and health care for patients in Ontario and internationally.

3. Research Plan

Objectives:

1. To develop a registry of patients undergoing FDG PET for the assessment of myocardial viability
2. To determine the upstream and downstream resource utilization (diagnostic imaging and revascularization) in patients undergoing FDG PET
3. To determine the outcome of patients undergoing PET imaging and relate this outcome to the severity of the abnormalities detected.
4. To determine the impact of FDG PET parameters on outcome measures compared to other clinical parameters.

Methods: Consent will be obtained from all eligible subjects. Data will be collected in a prospective manner to evaluate patients, who meet inclusion criteria, undergoing cardiac PET imaging. Physicians in Ontario will be notified via the Ontario Medical association (OMA)and Cardiovascular Care Network that FDG PET viability imaging is clinically available for appropriate patients through the provincial registry. The participating registry sites as well as indications for FDG PET viability imaging will be circulated.

Health Canada requires that all patients undergoing imaging with positron emitting radiopharmaceuticals (PERs) must partake in a research protocol, therefore for those patients who do not wish to participate in the CADRE study, a second consent is provided for the collection of baseline safety data only, ie imaging parameters, tracer dose and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic left ventricular dysfunction in the moderate to severe range (previous assessment of ventricular function with left ventricular ejection fraction (LVEF) approximately 35%
* Patients will be possible candidates for revascularization if sufficient viable myocardium is identified or considered for heart transplantation if there is no viable myocardium
* Patients with New York Heart Association (NYHA) or Canadian Cardiovascular Society (CCS) Class II - IV symptoms despite maximal medical therapy.

Exclusion Criteria:

* Under 18 years of age
* Pregnant or lactating females
* Already known to be ineligible for further revascularization or cardiac transplantation
* Unable to lie supine for imaging with PET
* Unable to take insulin (eg. severe hypokalemia)
* Failure to obtain informed consent
* Claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for cardiac FDG PET viability imaging
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2007-04; Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the composite clinical endpoint of cardiac death, myocardial infarction, transplantation, or re-hospitalization for unstable angina or heart failure. | 1 year

SECONDARY OUTCOMES:
Other outcomes will include death from any cause, revascularization, and downstream diagnostic utilization. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rob S. Beanlands, MD, FRCP C, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (4):
- Canada (4):
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No